CLINICAL TRIAL: NCT05137340
Title: Nasal Continuous Positive Airway Pressure Versus Non-invasive Positive Pressure Ventilation as Primary Support Before Minimally Invasive Surfactant Administration for Preterm Infants With NRDS
Brief Title: NIV-MISA-NRDS Trial: a Multicenter Study in China
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The trial was terminated early based on interim analysis results indicating futility. The decision was approved by the Data Safety Monitoring Committee (DSMC).
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: M2021378
Record Dates: First submitted 2021-11-28; First posted 2021-11-30 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-05

CONDITIONS: Minimal Invasive Surfactant Administration in Two Different Non-invasive Ventilation Modes to NRDS Infants
MeSH Terms: interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: A randomized, clinical, parallel-group study
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NCPAP group (Experimental): The ventilator parameter of NCPAP group are set with positive end expiratory pressure [PEEP] of 6cmH2O (adjustment range 6-8cmH2O) and FiO2 of 0.21-0.40, in order to maintain an oxygen saturation level of 90%-95%.
  Interventions: Other: Nasal continuous positive airway pressure
- NIPPV group (Active Comparator): NIPPV group are set with PEEP of 6cmH2O (adjustment range 6-8cmH2O), peak inspiratory pressure [PIP] of 15cmH2O (regulation range 15-20cmH2O), inspiratory time of 0.3s (regulation range 0.3-0.4s), respiratory rate of 30 times/min (regulation range 20-40 times/min) and FiO2 of 0.21-0.40.
  Interventions: Other: Non-invasive positive pressure ventilation

INTERVENTIONS:
Other: Nasal continuous positive airway pressure — Preterm infants with spontaneous breathing are stabilized on non-invasive respiratory support (PEEP of 6 cmH2O and FiO2≤0.40) in the delivery room and during admission to NICU, and then randomly selected to start NCPAP within 30 minutes of birth. Under NCPAP, the calf pulmonary surfactant will be administered via MISA method within 120 minutes after birth if infants are clinically diagnosed with RDS.
  Arms: NCPAP group
Other: Non-invasive positive pressure ventilation — Preterm infants with spontaneous breathing are stabilized on non-invasive respiratory support (PEEP of 6 cmH2O and FiO2≤0.40) in the delivery room and during admission to NICU, and then randomly selected to start NIPPV within 30 minutes of birth. Under NIPPV, the calf pulmonary surfactant will be administered via MISA method within 120 minutes after birth if infants are clinically diagnosed with RDS.
  Arms: NIPPV group

SUMMARY:
BACKGROUND Non-invasive ventilation (NIV) treatment have been developed to minimize lung damage and to avoid invasive mechanical ventilation (IMV) in preterm infants, especially in those with gestational age less than 30 weeks. Our hypothesis is that for preterm infants less than 30 weeks with potential to develop neonatal respiratory distress syndrome (NRDS), nasal continuous positive airway pressure (NCPAP) is non-inferior to the nasal intermittent positive pressure ventilation (NIPPV) as primary respiratory support before minimal invasive surfactant administration (MISA).

DESIGN, SETTING, AND PARTICIPANTS The NIV-MISA-NRDS trial is planned as an unblinded, multicenter, randomized, non-inferiority trial at 11 tertiary care neonatal intensive care units in China. Eligible infants are preterm infants of 24 to 29+6 weeks' gestational age who have spontaneous breaths at birth and require primary NIV support for NRDS in the first 2 h of life. Infants are randomized 1:1 to treatment with either NCPAP or NIPPV once admitted into neonatal intensive care unit (NICU). If the patient with progressively aggravates respiratory distress and clinically diagnose as NRDS, pulmonary surfactant will be supplemented by minimal invasive surfactant administration (MISA) in the first 2 hours .

MAIN OUTCOMES AND MEASURES The primary outcome is NIV treatment failure within 72 hours after birth, as determined by objective oxygenation, blood gas, and apnea criteria, or the need for intubation and mechanical ventilation. Secondary outcomes mainly include the incidence of complications during hospitalization . With a specified noninferiority margin of 10%, using a two-sided 95% CI and 80% power, the study requires 480 infants per group (total 960 infants in the study).

DETAILED DESCRIPTION:
The ventilator parameter of NCPAP group are set with positive end expiratory pressure [PEEP] of 6cmH2O (adjustment range 6-8cmH2O) and FiO2 of 0.21-0.40, in order to maintain an oxygen saturation level of 90%-95%.

NIPPV group are set with PEEP of 6cmH2O (adjustment range 6-8cmH2O), peak inspiratory pressure [PIP] of 15cmH2O (regulation range 15-20cmH2O), inspiratory time of 0.3s (regulation range 0.3-0.4s), respiratory rate of 30 times/min (regulation range 20-40 times/min) and FiO2 of 0.21-0.40.

ELIGIBILITY:
Inclusion Criteria

Infants who meet all of the following criteria will be included:

1. Infants of 24 to 29+6 weeks GA.
2. Infants with spontaneous breathing and signs of respiratory distress will receive non-invasive respiratory support (PEEP of 6 cmH2O and fraction of inspired oxygen[FiO2]≤0.40) immediately after birth in the delivery room and during transfer to NICU. Once the infant is settled down in the incubator, and the ventilation support of NCPAP or NIPPV by ventilator in NICU will by started according to the randomization of protocol.
3. Under NCPAP or NIPPV, the surfactant will be administered via MISA approach within 120 minutes after birth if the infant required FiO2>0.3 for transcutaneous oxygen saturation [SpO2]>85%, or Silverman Anderson Score [SAS] >5 points or SAS increasing >2 points per hour.
4. Parental consent will be obtained for all participants.

Exclusion Criteria

Infants who meet any of the following criteria will be excluded:

1. Infants who have been intubated prior to pulmonary surfactant administration due to postnatal resuscitation or other reasons.
2. Infants with obvious malformations affecting respiratory function.
3. Infants who have been transferred out to other hospitals for surgery or died for other complications with uncompleted data.
4. Infants who have participated in other interventional researches.

Ages: 30 Minutes to 4 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 312 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2025-02-01 (Actual); Study Completion 2025-03-10 (Actual)

PRIMARY OUTCOMES:
NIV treatment failure within the first 72 hours of life | From enrollment to the first 72 hours of life
  The failure of non-invasive nasal respiratory support(NIPPV or NCPAP) within the first 72 hours of life

SECONDARY OUTCOMES:
NIV treatment failure within 7days after birth | From enrollment to 7days after birth
  The failure of non-invasive nasal respiratory support(NIPPV or NCPAP) within 7days after birth
Rate of pneumothorax | Through study completion and up to corrected three months
  Rate of pneumothorax
Rate of pulmonary hemorrhage | Through study completion and up to corrected three months
  Rate of pulmonary hemorrhage
Rate of hemodynamically significant patent ductus arteriosus (hsPDA) | Through study completion and up to corrected three months
  Rate of hemodynamically significant patent ductus arteriosus (hsPDA)
Rate of intraventricular hemorrhages (IVH, grade III or Ⅳ) | Through study completion and up to corrected three months
  Rate of intraventricular hemorrhages (IVH, grade III or Ⅳ)
Rate of periventricular leukomalacia | Through study completion and up to corrected three months
  Rate of periventricular leukomalacia
Rate of late-onset sepsis | Through study completion and up to corrected three months
  Rate of late-onset sepsis
Rate of bronchopulmonary dysplasia (BPD) | At 36 weeks PMA
  Rate of bronchopulmonary dysplasia (BPD)
Rate of necrotizing enterocolitis (NEC) | Through study completion and up to corrected three months
  Rate of necrotizing enterocolitis (NEC)
Rate of retinopathy of prematurity (ROP) | Through study completion and up to corrected three months
  Rate of retinopathy of prematurity (ROP)
Duration of non-invasive ventilation, IMV, and supplemental oxygen | Through study completion and up to corrected three months
  Duration of non-invasive ventilation, duration of IMV, and days on supplemental oxygen
Length of hospital stay | From enrollment to the end of treatment at an average of 8 weeks
  Length of hospital stay
Required>1 doses of surfactant | From enrollment to 5 days after birth
  rate of required>1 doses of surfactant
In-hospital mortality | Through study completion and up to corrected three months
  In-hospital mortality
Pneumonia | Through study completion and up to corrected three months
  rate of pneumonia
Persistent pulmonary hypertension of newborn | Through study completion and up to corrected three months
  rate of persistent pulmonary hypertension of newborn

CONTACTS AND LOCATIONS:
Overall Officials: Xiaomei Tong, Tong,, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Li J, Zeng L, Gao Y, Zhao W, Han T, Tong X. A multicenter, randomized controlled, non-inferiority trial, comparing nasal continuous positive airway pressure with nasal intermittent positive pressure ventilation as primary support before minimally invasive surfactant administration for preterm infants with respiratory distress syndrome (the NIV-MISA-RDS trial): Study protocol. Front Pediatr. 2022 Jul 29;10:968462. doi: 10.3389/fped.2022.968462. eCollection 2022. PMID 35967549